CLINICAL TRIAL: NCT05708040
Title: Open-label, Randomized, Controlled Clinical Trial to Evaluate the Efficacy of the Smart Insulin Pen Associated With a Continuous Glucose Monitoring System Compared to a Closed Loop System in Patients With Type 1 Diabetes (EBIACE-1)
Brief Title: Clinical Trial to Evaluate the Efficacy of the Smart Insulin Pen Compared to a Closed Loop System in Patients With Type 1 Diabetes (EBIACE-1)
Acronym: EBIACE-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 189/22
Record Dates: First submitted 2023-01-12; First posted 2023-02-01 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed loop system (Active Comparator): Minimed 780G (Medtronic)
  Interventions: Device: InPen Medtronic
- SmartPen (Experimental): InPen (Medtronic)
  Interventions: Device: Minimed 780G system

INTERVENTIONS:
Device: InPen Medtronic — Patients with DM1 ≥ 18 years of age who initiate Inpen system.
  Arms: Closed loop system
Device: Minimed 780G system — Patients with DM1 ≥ 18 years of age who initiate Minimed 780G system.
  Arms: SmartPen

SUMMARY:
Analysis of glycemic control, frequency of hypoglycemia, glycemic variability, patient satisfaction and patient-perceived quality of life in patients with type 1 diabetes mellitus and continuous real-time glucose monitoring, the use of a smart pen compared to a closed loop system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for DM1 according to ADA
* Candidates for both systems (closed loop or smart insulin pen) for their usual healthcare team.
* Acceptance of participation in the study and signing of the informed consent

Exclusion Criteria:

* Gestation
* Institutionalization, serious or terminal illness or renal replacement therapy.
* Inability to undertake the training and / or acquire the degree of knowledge to use both systems
* Refusal to participate in the study or to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Time in Range | 12 months
  To assess the difference on the glycemic control expressed as time in range (% of time between 70-180 mg/dl of interstitial glucose).

SECONDARY OUTCOMES:
A1c levels | 12 months
  To assess the differences in serum A1c levels (%)
Time below range | 12 months
  To assess the difference on the glycemic control expressed as time in below range (% of time < 70 mg/dl of interstitial glucose).
Time above range | 12 months
  To assess the difference on the glycemic control expressed as time in above range (% of time >180 mg/dl of interstitial glucose).
Health-Related Quality of Life in Patients with Type 1 Diabetes | 12 months
  Assess health-related quality of life in patients with type 1 diabetes (by ViDa1 questionnaire).ViDa1 questionnaire has four-dimensional structure: Interference of diabetes in everyday life, Self-care, Well-being, and Worry about the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lía Nattero-Chávez, MD.PhD, Principal Investigator — Hospital Ramón y CajaDiabetes, Obesity and Human Reproduction Research Group, Department of Endocrinology and Nutrition, Hospital Universitario Ramón y Cajal, Universidad de Alcalá, Instituto Ramón y Cajal de Investigación Sanitaria (IRYCIS)
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain